CLINICAL TRIAL: NCT04677179
Title: An Adaptive Phase 2, Randomized, Double Blind, Placebo Controlled Study of LY3471851 (NKTR 358) in Patients With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study of LY3471851 in Adult Participants With Moderately to Severely Active Ulcerative Colitis (UC)
Acronym: INSTRUCT-UC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to enrollment futility.
Sponsor: Nektar Therapeutics (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17287; J1P-MC-KFAH (Other: Eli Lilly and Company); 2020-003017-35 (EudraCT Number)
Record Dates: First submitted 2020-12-08; First posted 2020-12-21 (Actual); Results first posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Colitis, Ulcerative
Keywords: T regulatory cells (Tregs); Interleukin 2; Interleukin-2
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High dose LY3471851 (Experimental): Participants received a subcutaneous injection of high dose LY3471851 every 2 weeks from weeks 0 to 12. Week 12 responders entered the maintenance period and continued with the same treatment. Week 12 non-responders entered the extension period where they received subcutaneous injection of high dose LY3471851 every 2 weeks up to week 50. At week 26, extension period non-responders were discontinued from treatment. Post-treatment, participants entered follow-up period and were observed for 6 weeks for safety.
  Interventions: Drug: LY3471851
- Low dose LY3471851 (Experimental): Participants received a subcutaneous injection of low dose LY3471851 every 2 weeks from weeks 0 to 12. Week 12 responders entered the maintenance period and continued with the same treatment. Week 12 non-responders entered the extension period where they received subcutaneous injection of high dose LY3471851 every 2 weeks up to week 50. At week 26, extension period non-responders were discontinued from treatment. Post-treatment, participants entered follow-up period and were observed for 6 weeks for safety.
  Interventions: Drug: LY3471851
- Placebo (Placebo Comparator): Participants received a subcutaneous injection of placebo every 2 weeks from weeks 0 to 12. Week 12 responders entered the maintenance period and continued with the same treatment. Week 12 non-responders entered the extension period where they received subcutaneous injection of high dose LY3471851 every 2 weeks up to week 50. At week 26, extension period non-responders were discontinued from treatment. Post-treatment, participants entered follow-up period and were observed for 6 weeks for safety.
  Interventions: Drug: LY3471851; Drug: Placebo

INTERVENTIONS:
Drug: LY3471851 — administered SC
  Other Names: NKTR-358
Drug: Placebo — administered SC
  Arms: Placebo

SUMMARY:
The reason for this study is to determine if the study drug LY3471851 is safe and effective in adult participants with active ulcerative colitis (UC). The study treatment will last about 52 weeks.

DETAILED DESCRIPTION:
In stage 1, two doses (high and low) of LY3471851 will be compared to placebo. In stage 2, up to two additional doses (to be confirmed) of LY3471851 will be compared to placebo.

LY3471851 (NKTR-358) is a potential first-in-class therapeutic that may address an underlying immune system imbalance in people with many autoimmune conditions. It targets the interleukin (IL-2) receptor complex in the body in order to stimulate proliferation of inhibitory immune cells known as regulatory T cells. By activating these cells, LY3471851 may act to bring the immune system back into balance.

ELIGIBILITY:
Inclusion Criteria:

* Have moderately to severely active ulcerative colitis (UC) as defined by a modified Mayo score (MMS) of 4 to 9 with an endoscopic subscore (ES) ≥2, with endoscopy performed within 14 days before baseline.
* Have evidence of UC extending proximal to the rectum (with ≥15 centimeters (cm) of involved colon).
* Have up-to-date colorectal cancer surveillance performed according to local standard.
* Participants are either one of the following:
* Have failed conventional treatments including inability to tolerate oral or intravenous corticosteroids or immunomodulators (6-mercaptopurine or azathioprine or methotrexate), or history of corticosteroid dependence (an inability to successfully taper corticosteroids without return of UC) and neither failed or demonstrated intolerance to advanced therapy (eg, tumor necrosis factor (TNF) antagonists, anti-integrin therapies, anti-IL12/23p40 therapies, Janus kinase (JAK) inhibitor) OR,
* Have failed advanced therapies such as treatment with 1 or more advance therapies (eg, tumor necrosis factor [TNF] antagonists, anti-integrin therapies, anti-IL12/23p40 therapies, Janus kinase [JAK] inhibitor) at doses approved for the treatment of UC with documented history of failure to respond to or tolerate such treatment.
* Have had an established diagnosis of UC of ≥3 months in duration before baseline which includes endoscopic evidence of UC and a histopathology report that supports a diagnosis of UC. Supportive endoscopy and histopathology reports must be available in the source documents.
* Women of child-bearing potential (WOCBP) must test negative for pregnancy as indicated by a negative serum pregnancy test at the screening visit followed by a negative urine pregnancy test within 24 hours prior to first exposure to study drug.

Exclusion Criteria:

* Have been diagnosed with indeterminant colitis, proctitis (colitis limited to the rectum only; less than 15 centimeter (cm) from the anal verge or Crohn's disease.
* Have received any of the following for treatment of UC: cyclosporine, tacrolimus, mycophenolate mofetil or thalidomide within 2 weeks of screening, rectally administered corticosteroids or 5-aminosalicylic acid treatments within 2 weeks of screening.
* Have had or will need abdominal surgery for UC (for example, subtotal colectomy).
* Have failed 3 or more classes of advanced therapies approved for treatment of UC (eg, tumor necrosis factor [TNF] antagonists, anti-integrin therapies, anti-IL12/23p40 therapies, Janus kinase [JAK] inhibitor).
* Have evidence of toxic megacolon, intra-abdominal abscess, or stricture/stenosis within the small bowel or colon.
* Have any history or evidence of cancer of the gastrointestinal tract
* Have myocardial infarction, unstable ischemic heart disease, stroke or heart failure within 12 months prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (116):
- United States (7):
  - Dedicated Clinical Research, Litchfield Park, Arizona
  - I.H.S. Health, LLC, Kissimmee, Florida
  - Gastroenterology Associates of Pensacola, PA, Pensacola, Florida
  - Atlantic Digestive Health Institute, Morristown, New Jersey
  - Biopharma Informatic, LLC, Houston, Texas
  - Southern Star Research Institute, LLC, San Antonio, Texas
  - Care Access Research - Ogden, Ogden, Utah
- Argentina (4):
  - DOM- Centro de Reumatologia, CABA, Buenos Aires
  - Centro de Educación Médica e Investigaciones Clínicas "Norberto Quirno" CEMIC, CABA, Buenos Aires
  - Mautalen Salud e Investigacion-Centro de Osteopatías Médicas, Ciudad Autonoma de Buenos Air, Buenos Aires
  - Centro Médico Privado de Reumatología, San Miguel de Tucumán
- Australia (4):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Paratus Clinical Research Brisbane, Albion, Queensland
  - Mater Adult Hospital Brisbane, South Brisbane, Queensland
  - St. Vincent's Hospital, Fitzroy, Victoria
- Belgium (3):
  - Université Libre de Bruxelles - Hôpital Erasme, Brussels, Bruxelles-Capitale, Région de
  - Centre Hospitalier de Wallonie Picarde - Site Notre Dame, Tournai, Wallonne, Région
  - AZ Maria Middelares, Ghent
- Brazil (8):
  - Chronos Pesquisa Clínica, Brasília, Federal District
  - Nucleo de Pesquisa Clínica do Rio Grande do Sul-NPCRS, Porto Alegre, Rio Grande do Sul
  - Upeclin - Unidade de Pesquisa Clínica da Faculdade de Medicina de Botucatu - UNESP, Botucatu, São Paulo
  - HMCP - Hospital e Maternidade Celso Pierro - PUC-Campinas, Campinas, São Paulo
  - Pesquisare, Santo André, São Paulo
  - CEMEC - Centro Multidisciplinar de Estudos Clinicos EPP Ltda, São Bernardo do Campo, São Paulo
  - Instituto de Assistencia Medica ao Servidor Publico Estudo Estadual, São Paulo, São Paulo
  - Hepatogastro, São Paulo
- Canada (4):
  - Gastroenterology and internal medicine research institute, Edmonton, Alberta
  - Gastroenterology Research, Nova Scotia Health Authority, Halifax, Nova Scotia
  - CISSS de la Montérégie - Centre Hôpital Charles-Le Moyne, Greenfield Park, Quebec
  - McGill University, Montreal, Quebec
- China (9):
  - The First Affiliated Hospital of Anhui Medical University, HefeiCity, Anhui
  - First affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hosp Tongji Med Col Huazhong Univ of Sci & Tech, Wuhan, Hubei
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Taian City Central Hospital, Taian, Shandong
  - Shanghai Jiaotong University School of Medicine Ruijin Hospital, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
- Czechia (5):
  - A-Shine, Pilsen, Plzeň-město
  - MUDr. Gregar, s.r.o., Olomouc
  - PreventaMed, s.r.o., Olomouc
  - I. Interni klinika FN Plzen, Plzen-Lochotin
  - Nemocnice Slaný, Slaný
- France (2):
  - CHU De Grenoble Hopital Albert Michallon, Grenoble
  - Centre Hospitalier de Mont de Marsan, Mont-de-Marsan
- Georgia (2):
  - Acad. F. Todua Medical Center - Research Institute of Clinical Medicine, Tbilisi
  - Medical Center: Medinvestment, Tbilisi
- Hungary (4):
  - Clinexpert SMO, Budapest
  - Óbudai Egészségügyi Centrum, Budapest
  - Bugát Pál Kórház, Gyöngyös
  - CLINFAN Szolgáltató Kft, Szekszárd
- India (8):
  - Shree Giriraj Multispeciality Hospital, Rajkot, Gujarat
  - Gujarat Hospital - Gastro and Vascular Centre, Surat, Gujarat
  - Kingsway Hospital, Nagpur, Maharashtra
  - Midas Multispeciality Hospital Pvt.Ltd., Nagpur, Maharashtra
  - SR Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - Apollo Speciality Hospital - Teynampet, Chennai, Tamil Nadu
  - Postgraduate Institute of Medical Education & Research, Chandigarh
  - Gandhi Hospital, Telangana
- Israel (3):
  - Soroka Medical Center, Beersheba
  - Galilee Medical Center - Internal A, Nahariya
  - Kaplan Medical Center, Rehovot
- Japan (13):
  - Fukuoka University Chikushi Hospital, Chikushino-shi, Fukuoka
  - Tokushukai Sapporo Tokushukai Hospital, Sapporo, Hokkaido
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Sai Gastroenterologist Proctology, Fujiidera, Osaka
  - Infusion Clinic, Osaka, Osaka
  - Matsuda Hospital, Hamamatsu, Shizuoka
  - Showa University Koto Toyosu Hospital, Koto-ku, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku-ku, Tokyo-To
  - Fukuoka University Hospital, Fukuoka
  - Sameshima Hospital, Kagoshima
  - Toyama Prefectural Central Hospital, Toyama
  - Yamagata University Hospital, Yamagata
- Pauls Stradins Clinical Univeristy Hospital, Riga, Rīga, Latvia
- Poland (4):
  - NZOZ Vivamed, Warsaw, Masovian Voivodeship
  - Szpital Miejski Sw. Jana Pawla II, Elblag
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - ETG Zamość, Zamość
- Romania (6):
  - SC Pelican SRL, Oradea, Bihor County
  - SC Med Life SA, Bucharest
  - SC Centrul Medical Sana SRL, Bucharest
  - Spital Clinic Colentina, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj, Cluj-Napoca
  - S.C. Materna Care S.R.L., Timișoara
- Russia (7):
  - Olla-Med, Moscow, Moscow
  - Novosibirski Gastrocenter, Novosibirsk, Novosibirsk Oblast
  - Rostov State Medical University, Rostov-on-Don, Rostov Oblast
  - Open Joint Stock Company Clinical and Diagnostic Center Euromedservice, Moscow
  - The University Clinic of OSMU, Omsk
  - SPb SBIH "City Mariinskaya Hospital", Saint Petersburg
  - GOU VPO St-Petersburg SMA n/a Mechnikov Fed. Agen of Health, Saint Petersburg
- Slovakia (2):
  - FNsP FDRoosevelta Banska Bystrica, Banská Bystrica
  - ENDOMED s.r.o., Košice
- South Korea (5):
  - Yonsei University Wonju Severance Christian Hospital, Gangwon-do, Gangwon-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Samsung Medical Center, Seoul, Korea
  - Seoul St. Mary's Hospital, Seoul, Korea
  - Inje University Haeundae Paik Hospital, Busan
- Ukraine (10):
  - Medical Center of Limited Liability Company "Medical Center "Consilium Medical", Kiev, Kyiv Oblast
  - Lviv Railway Clinical Hospital, Lviv, Lviv Oblast
  - Lviv Regional Endocrinology Dispensary, Lviv, Lviv Oblast
  - Medical Center of LLC Medical Center Clinic of Family Medicine, Dnipro
  - International Institute of Clinical Trials LLC, Kyiv
  - Communal Enterprise "Odesa Regional Clinical Hospital", Odesa
  - A. Novak Transcarpathian Regional Clinical Hospital, Uzhhorod
  - CCH #1 Vinnytsia M.I. Pyrogov NMU Ch of Propaedeutics of IM, Vinnytsia
  - Vinnytsia War Veterans Regional Clinical Hospital, Vinnytsia
  - Diacenter LLC, Zaporizhzhia
- United Kingdom (5):
  - Royal Derby Hospital, Derby, Derbyshire
  - Whipps Cross University Hospital, Leytonstone, London
  - Guys/St. Thomas Hospital, London, Surrey
  - St. George's Hospital, London
  - York Hospital, York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3471851 in Adult Participants With Moderately to Severely Active Ulcerative Colitis (UC) ( INSTRUCT-UC ) — https://trials.lillytrialguide.com/en-US/trial/V3FQqG8aJfjj6JtJ60xFt

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of:
  * a 12-week induction treatment period: participants randomly received either high dose LY3471851 or low dose LY3471851 or placebo.
  * a 40-week maintenance/extension treatment period (final dose at week 50 and study assessments at week 52)
  * (i) Week 12 responders enter the maintenance period where they continued to receive the same treatment to which they were randomly assigned.
  (Continued..)
Pre-assignment Details: * (ii) Week 12 non-responders enter the extension period where they received high dose LY3471851. At week 26, those who responded to treatment continued with the same treatment, while non-responders discontinued and entered follow-up.
  * a 6-week post-treatment follow-up period: Following treatment completion or discontinuation, participants entered the follow-up period and were observed for safety. No treatments were administered.
Groups:
- High Dose LY3471851 (Induction Treatment Period): Participants received a subcutaneous injection of high dose LY3471851 every 2 weeks from weeks 0 to 12.
- Low Dose LY3471851 (Induction Treatment Period): Participants received a subcutaneous injection of low dose LY3471851 every 2 weeks from weeks 0 to 12.
- Placebo (Induction Treatment Period): Participants received a subcutaneous injection of placebo every 2 weeks from weeks 0 to 12.
- High Dose LY3471851 (Maintenance Treatment Period): Week 12 responders from the high dose LY3471851 induction treatment period arm entered the maintenance period and continued with the same treatment.
- Low Dose LY3471851 (Maintenance Treatment Period): Week 12 responders from the low dose LY3471851 induction treatment period arm entered the maintenance period and continued with the same treatment.
- Placebo (Maintenance Treatment Period): Week 12 responders from the placebo induction treatment period arm entered the maintenance period and continued with the same treatment.
- High Dose LY3471851 (Extension Treatment Period): Week 12 non-responders entered the extension period where they received subcutaneous injection of high dose LY3471851 every 2 weeks up to week 50. At week 26, extension period non-responders were discontinued from treatment.
- High Dose LY3471851 (Post-Treatment Follow-up Period): Participants randomised to high dose LY3471851 arm entered follow-up period from induction or maintenance, or extension periods and were observed for 6 weeks for safety. No treatments were administered.
- Low Dose LY3471851 (Post-Treatment Follow-up Period): Participants randomised to low dose LY3471851 arm entered follow-up period from induction or maintenance, or extension periods and were observed for 6 weeks for safety. No treatments were administered.
- Placebo (Post-Treatment Follow-up Period): Participants randomised to placebo arm entered follow-up period from induction or maintenance, or extension periods and were observed for 6 weeks for safety. No treatments were administered.
Period: Induction Treatment Period
Arm/Group | High Dose LY3471851 (Induction Treatment Period) | Low Dose LY3471851 (Induction Treatment Period) | Placebo (Induction Treatment Period) | High Dose LY3471851 (Maintenance Treatment Period) | Low Dose LY3471851 (Maintenance Treatment Period) | Placebo (Maintenance Treatment Period) | High Dose LY3471851 (Extension Treatment Period) | High Dose LY3471851 (Post-Treatment Follow-up Period) | Low Dose LY3471851 (Post-Treatment Follow-up Period) | Placebo (Post-Treatment Follow-up Period)
Started | 32 | 35 | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 32 | 35 | 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 19 | 22 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 13 | 13 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 7 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Treatment Period
Arm/Group | High Dose LY3471851 (Induction Treatment Period) | Low Dose LY3471851 (Induction Treatment Period) | Placebo (Induction Treatment Period) | High Dose LY3471851 (Maintenance Treatment Period) | Low Dose LY3471851 (Maintenance Treatment Period) | Placebo (Maintenance Treatment Period) | High Dose LY3471851 (Extension Treatment Period) | High Dose LY3471851 (Post-Treatment Follow-up Period) | Low Dose LY3471851 (Post-Treatment Follow-up Period) | Placebo (Post-Treatment Follow-up Period)
Started | 0 (Induction treatment period arm.) | 0 (Induction treatment period arm.) | 0 (Induction treatment period arm.) | 8 (Only week 12 induction treatment responders entered the maintenance treatment period.) | 10 (Only week 12 induction treatment responders entered the maintenance treatment period.) | 5 (Only week 12 induction treatment responders entered the maintenance treatment period.) | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 8 | 10 | 5 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 7 | 9 | 5 | 0 | 0 | 0 | 0
Period: Extension Treatment Period
Arm/Group | High Dose LY3471851 (Induction Treatment Period) | Low Dose LY3471851 (Induction Treatment Period) | Placebo (Induction Treatment Period) | High Dose LY3471851 (Maintenance Treatment Period) | Low Dose LY3471851 (Maintenance Treatment Period) | Placebo (Maintenance Treatment Period) | High Dose LY3471851 (Extension Treatment Period) | High Dose LY3471851 (Post-Treatment Follow-up Period) | Low Dose LY3471851 (Post-Treatment Follow-up Period) | Placebo (Post-Treatment Follow-up Period)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 26 (Only week 12 induction treatment non-responders entered the extension treatment period.) | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 0 | 0 | 0
Period: Post-Treatment Follow-up Period
Arm/Group | High Dose LY3471851 (Induction Treatment Period) | Low Dose LY3471851 (Induction Treatment Period) | Placebo (Induction Treatment Period) | High Dose LY3471851 (Maintenance Treatment Period) | Low Dose LY3471851 (Maintenance Treatment Period) | Placebo (Maintenance Treatment Period) | High Dose LY3471851 (Extension Treatment Period) | High Dose LY3471851 (Post-Treatment Follow-up Period) | Low Dose LY3471851 (Post-Treatment Follow-up Period) | Placebo (Post-Treatment Follow-up Period)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 25 (Participants entered the post-treatment follow-up period from induction or maintenance, or extension treatment periods.) | 30 (Participants entered the post-treatment follow-up period from induction or maintenance, or extension treatment periods.) | 11 (Participants entered the post-treatment follow-up period from induction or maintenance, or extension treatment periods.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 25 | 30 | 11
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 26 | 11

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose LY3471851 (Induction Treatment Period) | Low Dose LY3471851 (Induction Treatment Period) | Placebo (Induction Treatment Period) | Total
Number analyzed (Participants) | 32 | 35 | 14 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (12.5) | 44.5 (13.8) | 45.7 (15.2) | 42.6 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 6 | 25
  Male | 22 | 26 | 8 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 4 | 2 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 2
  White | 25 | 31 | 12 | 68
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: All randomized participants with non-missing region of enrollment data.
  Participants
    Argentina: number analyzed (Participants) | 31 | 35 | 14 | 80
    Argentina | 2 | 1 | 1 | 4
    Australia: number analyzed (Participants) | 31 | 35 | 14 | 80
    Australia | 0 | 1 | 0 | 1
    Belgium: number analyzed (Participants) | 31 | 35 | 14 | 80
    Belgium | 0 | 0 | 1 | 1
    Czechia: number analyzed (Participants) | 31 | 35 | 14 | 80
    Czechia | 2 | 4 | 0 | 6
    Hungary: number analyzed (Participants) | 31 | 35 | 14 | 80
    Hungary | 3 | 3 | 0 | 6
    Japan: number analyzed (Participants) | 31 | 35 | 14 | 80
    Japan | 3 | 1 | 1 | 5
    South Korea: number analyzed (Participants) | 31 | 35 | 14 | 80
    South Korea | 1 | 3 | 1 | 5
    Latvia: number analyzed (Participants) | 31 | 35 | 14 | 80
    Latvia | 2 | 3 | 0 | 5
    Poland: number analyzed (Participants) | 31 | 35 | 14 | 80
    Poland | 2 | 2 | 1 | 5
    Russia: number analyzed (Participants) | 31 | 35 | 14 | 80
    Russia | 5 | 5 | 3 | 13
    Slovakia: number analyzed (Participants) | 31 | 35 | 14 | 80
    Slovakia | 1 | 1 | 1 | 3
    Ukraine: number analyzed (Participants) | 31 | 35 | 14 | 80
    Ukraine | 7 | 7 | 4 | 18
    United States: number analyzed (Participants) | 31 | 35 | 14 | 80
    United States | 3 | 4 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Clinical Remission at Week 12
Description: Clinical remission is defined as achieving a Modified Mayo Score (MMS) sub-score for rectal bleeding=0, stool frequency=0, or stool frequency=1 with ≥ 1 point decrease from baseline, and endoscopy=0 or 1 (excluding friability). The MMS is a scoring system for assessment of UC and is composed of sub-scores of stool frequency (range: 0 to 3, where 0=normal number of stools, 3=5 or more stools more than normal), endoscopy (range: 0 to 3, where 0=normal or inactive disease, 3=severe disease [spontaneous bleeding, ulceration]), rectal bleeding (range: 0 to 3, where 0=no blood seen, 3=blood alone passed). Total MMS score is sum of all sub-scores and ranges from 0 to 9, with higher scores indicating higher disease activity.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study drug and had MMS data at week 12.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Induction Treatment Period) | Low Dose LY3471851 (Induction Treatment Period) | High Dose LY3471851 (Induction Treatment Period)
Number analyzed (Participants) | 14 | 28 | 29
percentage of participants | 14.3 [0 to 32.6] | 7.1 [0 to 16.7] | 17.2 [3.5 to 31]
Statistical Analysis 1: Comparison: Placebo (Induction Treatment Period) vs Low Dose LY3471851 (Induction Treatment Period); Test type: Superiority; p = 0.750, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.57, 95% CI 2-sided [0.03 to 11.32]
Statistical Analysis 2: Comparison: Placebo (Induction Treatment Period) vs High Dose LY3471851 (Induction Treatment Period); Test type: Superiority; p = 0.838, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.10 to 6.21]

2. Secondary Outcome: Percentage of Participants Who Achieved Clinical Response at Week 12
Description: Clinical response is defined as a decrease in the MMS of ≥2 points and ≥30% decrease from baseline, and a decrease of ≥1 point in the rectal bleeding sub-score from baseline or a rectal bleeding score of 0 or 1. The MMS is a scoring system for assessment of UC and is composed of sub-scores of stool frequency (range: 0 to 3, where 0=normal number of stools, 3=5 or more stools more than normal), endoscopy (range: 0 to 3, where 0=normal or inactive disease, 3=severe disease [spontaneous bleeding, ulceration]), rectal bleeding (range: 0 to 3, where 0=no blood seen, 3=blood alone passed). Total MMS score is sum of all sub-scores and ranges from 0 to 9, with higher scores indicating higher disease activity.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study drug and had MMS data at week 12.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Induction Treatment Period) | Low Dose LY3471851 (Induction Treatment Period) | High Dose LY3471851 (Induction Treatment Period)
Number analyzed (Participants) | 14 | 28 | 29
percentage of participants | 35.7 [10.6 to 60.8] | 39.3 [21.2 to 57.4] | 41.4 [23.5 to 59.3]
Statistical Analysis 1: Comparison: Placebo (Induction Treatment Period) vs Low Dose LY3471851 (Induction Treatment Period); Test type: Superiority; p = 0.563, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.57, 95% CI 2-sided [0.10 to 3.30]
Statistical Analysis 2: Comparison: Placebo (Induction Treatment Period) vs High Dose LY3471851 (Induction Treatment Period); Test type: Superiority; p = 0.759, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.17 to 3.64]

3. Secondary Outcome: Percentage of Participants Who Achieved Endoscopic Remission at Week 12
Description: Endoscopic remission is defined as achieving a MMS sub-score for endoscopy=0 or 1 (excluding friability). The MMS is a scoring system for assessment of UC and is composed of sub-scores of stool frequency (range: 0 to 3, where 0=normal number of stools, 3=5 or more stools more than normal), endoscopy (range: 0 to 3, where 0=normal or inactive disease, 3=severe disease [spontaneous bleeding, ulceration]), rectal bleeding (range: 0 to 3, where 0=no blood seen, 3=blood alone passed). Total MMS score is sum of all sub-scores and ranges from 0 to 9, with higher scores indicating higher disease activity.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study drug and had MMS data at week 12.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Induction Treatment Period) | Low Dose LY3471851 (Induction Treatment Period) | High Dose LY3471851 (Induction Treatment Period)
Number analyzed (Participants) | 14 | 28 | 29
percentage of participants | 28.6 [4.9 to 52.2] | 14.3 [1.3 to 27.2] | 24.1 [8.6 to 39.7]
Statistical Analysis 1: Comparison: Placebo (Induction Treatment Period) vs Low Dose LY3471851 (Induction Treatment Period); Test type: Superiority; p = 0.163, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.18, 95% CI 2-sided [0.02 to 1.93]
Statistical Analysis 2: Comparison: Placebo (Induction Treatment Period) vs High Dose LY3471851 (Induction Treatment Period); Test type: Superiority; p = 0.439, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.11 to 2.77]

4. Secondary Outcome: Percentage of Participants Who Achieved Endoscopic Response at Week 12
Description: Endoscopic response is defined as a decrease of ≥1 point in the MMS endoscopy sub-score from baseline. The MMS is a scoring system for assessment of UC and is composed of sub-scores of stool frequency (range: 0 to 3, where 0=normal number of stools, 3=5 or more stools more than normal), endoscopy (range: 0 to 3, where 0=normal or inactive disease, 3=severe disease [spontaneous bleeding, ulceration]), rectal bleeding (range: 0 to 3, where 0=no blood seen, 3=blood alone passed). Total MMS score is sum of all sub-scores and ranges from 0 to 9, with higher scores indicating higher disease activity.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study drug and had MMS data at week 12.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Induction Treatment Period) | Low Dose LY3471851 (Induction Treatment Period) | High Dose LY3471851 (Induction Treatment Period)
Number analyzed (Participants) | 14 | 28 | 29
percentage of participants | 21.4 [0 to 42.9] | 32.1 [14.8 to 49.4] | 37.9 [20.3 to 55.6]
Statistical Analysis 1: Comparison: Placebo (Induction Treatment Period) vs Low Dose LY3471851 (Induction Treatment Period); Test type: Superiority; p = 0.821, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.17 to 9.88]
Statistical Analysis 2: Comparison: Placebo (Induction Treatment Period) vs High Dose LY3471851 (Induction Treatment Period); Test type: Superiority; p = 0.572, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.37 to 5.49]

5. Secondary Outcome: Percentage of Participants Who Achieved Symptomatic Remission at Week 12
Description: Symptomatic remission is defined as achieving a MMS sub-score for stool frequency=0, or stool frequency=1 with a decrease of ≥1 point from baseline, and rectal bleeding =0. The MMS is a scoring system for assessment of UC and is composed of sub-scores of stool frequency (range: 0 to 3, where 0=normal number of stools, 3=5 or more stools more than normal), endoscopy (range: 0 to 3, where 0=normal or inactive disease, 3=severe disease [spontaneous bleeding, ulceration]), rectal bleeding (range: 0 to 3, where 0=no blood seen, 3=blood alone passed). Total MMS score is sum of all sub-scores and ranges from 0 to 9, with higher scores indicating higher disease activity.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study drug and had MMS data at week 12.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Induction Treatment Period) | Low Dose LY3471851 (Induction Treatment Period) | High Dose LY3471851 (Induction Treatment Period)
Number analyzed (Participants) | 14 | 28 | 29
percentage of participants | 21.4 [0 to 42.9] | 32.1 [14.8 to 49.4] | 27.6 [11.3 to 43.9]
Statistical Analysis 1: Comparison: Placebo (Induction Treatment Period) vs Low Dose LY3471851 (Induction Treatment Period); Test type: Superiority; p = 0.886, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.14 to 10.16]
Statistical Analysis 2: Comparison: Placebo (Induction Treatment Period) vs High Dose LY3471851 (Induction Treatment Period); Test type: Superiority; p = 0.784, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.14 to 4.18]

6. Secondary Outcome: Percentage of Participants Who Achieved Symptomatic Response at Week 12
Description: Symptomatic response is defined as a ≥30% decrease from baseline in the composite clinical endpoint of the sum of MMS sub-scores of stool frequency and rectal bleeding. The MMS is a scoring system for assessment of UC and is composed of sub-scores of stool frequency (range: 0 to 3, where 0=normal number of stools, 3=5 or more stools more than normal), endoscopy (range: 0 to 3, where 0=normal or inactive disease, 3=severe disease [spontaneous bleeding, ulceration]), rectal bleeding (range: 0 to 3, where 0=no blood seen, 3=blood alone passed). Total MMS score is sum of all sub-scores and ranges from 0 to 9, with higher scores indicating higher disease activity.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study drug and had MMS data at week 12.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Induction Treatment Period) | Low Dose LY3471851 (Induction Treatment Period) | High Dose LY3471851 (Induction Treatment Period)
Number analyzed (Participants) | 14 | 28 | 29
percentage of participants | 42.9 [16.9 to 68.8] | 42.9 [24.5 to 61.2] | 44.8 [26.7 to 62.9]
Statistical Analysis 1: Comparison: Placebo (Induction Treatment Period) vs Low Dose LY3471851 (Induction Treatment Period); Test type: Superiority; p = 0.331, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.37, 95% CI 2-sided [0.06 to 2.43]
Statistical Analysis 2: Comparison: Placebo (Induction Treatment Period) vs High Dose LY3471851 (Induction Treatment Period); Test type: Superiority; p = 0.407, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.51, 95% CI 2-sided [0.10 to 2.52]

7. Secondary Outcome: Percentage of Participants Who Achieved Histologic Remission at Week 12
Description: Histologic Remission is defined as Geboes score <2 or subscores = 0 for Grade 2a, 2b, 3, 4, and 5. The Geboes score is a 7-item instrument used to identify histologic changes in UC. The 7 items are Grade 0: Architectural changes (0=No abnormality to 3=Severe diffuse or multifocal abnormalities); Grade 1: Chronic inflammatory infiltrate (0=No increase to 3=Marked increase); Grade 2A: lamina propria eosinophils (0=No increase to 3=Marked increase); Grade 2B: lamina propria neutrophils (0= No increase to 3=Marked increase); Grade 3: Neutrophils in epithelium (0=None to 3=>50% crypts involved); Grade 4: Crypt destruction(0=none to 3=Unequivocal crypt destruction),and Grade 5: Erosion or ulceration:(0=No erosion, ulceration or granulation to 4=Ulcer or granulation tissue). The grade with severe histological observation is considered the Geboes score and ranges from 0 to 4, with higher scores indicating severe disease.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study drug and had Geboes data at week 12.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Induction Treatment Period) | Low Dose LY3471851 (Induction Treatment Period) | High Dose LY3471851 (Induction Treatment Period)
Number analyzed (Participants) | 14 | 28 | 29
percentage of participants | 7.1 [0.0 to 20.6] | 7.1 [0.0 to 16.7] | 10.3 [0.0 to 21.4]
Statistical Analysis 1: Comparison: Placebo (Induction Treatment Period) vs Low Dose LY3471851 (Induction Treatment Period); Test type: Superiority; p = 0.564, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.50, 95% CI 2-sided [0.38 to 6.00]
Statistical Analysis 2: Comparison: Placebo (Induction Treatment Period) vs High Dose LY3471851 (Induction Treatment Period); Test type: Superiority; p = 0.681, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.51, 95% CI 2-sided [0.21 to 10.97]

8. Secondary Outcome: Percentage of Participants Who Achieved Histologic-Endoscopic Mucosal Healing (HEMH)
Description: HEMH is defined as Geboes score <2 AND endoscopic remission. Geboes score is a 7-item instrument used to identify histologic changes in UC. The 7-items are Grade 0: Architectural changes (0=No abnormality to 3=Severe diffuse or multifocal abnormalities); Grade 1: Chronic inflammatory infiltrate (0=No increase to 3=Marked increase); Grade 2A: lamina propria eosinophils (0=No increase to 3=Marked increase); Grade 2B: lamina propria neutrophils (0= No increase to 3=Marked increase); Grade 3: Neutrophils in epithelium (0=None to 3=>50% crypts involved); Grade 4: Crypt destruction(0=none to 3=Unequivocal crypt destruction),and Grade 5: Erosion or ulceration:(0=No erosion, ulceration or granulation to 4=Ulcer or granulation tissue). The grade with severe histological observation is considered the Geboes score and ranges from 0 to 4, with higher scores indicating severe disease. Endoscopic remission is defined as achieving a MMS sub-score for endoscopy=0 or 1 (excluding friability).
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study drug and had Geboes, MMS data at week 12.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Induction Treatment Period) | Low Dose LY3471851 (Induction Treatment Period) | High Dose LY3471851 (Induction Treatment Period)
Number analyzed (Participants) | 14 | 28 | 29
percentage of participants | 0 [0 to 0] | 3.6 [0 to 10.4] | 6.9 [0 to 16.1]
Statistical Analysis 1: Comparison: Placebo (Induction Treatment Period) vs Low Dose LY3471851 (Induction Treatment Period); Test type: Superiority; p = 0.317, Cochran-Mantel-Haenszel; Risk Difference (RD) = 3.6, 95% CI 2-sided [-3.3 to 10.4]
Statistical Analysis 2: Comparison: Placebo (Induction Treatment Period) vs High Dose LY3471851 (Induction Treatment Period); Test type: Superiority; p = 0.238, Cochran-Mantel-Haenszel; Risk Difference (RD) = 6.9, 95% CI 2-sided [-2.3 to 16.1]

9. Secondary Outcome: Change From Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) - Total Score
Description: IBDQ is a 32-item questionnaire that measures four aspects of participants' lives: symptoms directly related to the primary bowel disturbance (10 items), systemic symptoms (5 items), emotional function (12 items), and social function (5 items). Responses are graded on a 7-point Likert scale, where 7 denotes "not a problem at all" and 1 denotes "a very severe problem." The responses are summed to produce a total score ranging from 32 to 224, with higher score indicating a better quality of life. LS Mean was calculated using ANCOVA (analysis of covariance) model with treatment, baseline value, previous advanced therapy failure status (yes/no), baseline corticosteroid use (yes/no), baseline disease activity (MMS: [4 to 6] or [7 to 9]) and region (North America/Europe/Other) as fixed factors.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug and had IBDQ data at baseline, week 12.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo (Induction Treatment Period) | Low Dose LY3471851 (Induction Treatment Period) | High Dose LY3471851 (Induction Treatment Period)
Number analyzed (Participants) | 13 | 26 | 29
score on a scale | 26.71 (9.346) | 36.42 (7.640) | 25.76 (7.143)
Statistical Analysis 1: Comparison: Placebo (Induction Treatment Period) vs Low Dose LY3471851 (Induction Treatment Period); Test type: Superiority; p = 0.378, ANCOVA; LS Mean Difference = 9.71, 95% CI 2-sided [-12.17 to 31.60], Standard Error of Mean 10.935
Statistical Analysis 2: Comparison: Placebo (Induction Treatment Period) vs High Dose LY3471851 (Induction Treatment Period); Test type: Superiority; p = 0.928, ANCOVA; LS Mean Difference = -0.95, 95% CI 2-sided [-21.78 to 19.88], Standard Error of Mean 10.406

10. Secondary Outcome: Pharmacokinetics (PK): Trough Concentration of LY3471851 (Ctrough) at Week 12
Description: C-trough is the concentration of drug in the blood immediately before the next dose was administered.
Time Frame: Predose at week 12
Population: All participants who received at least 1 dose of LY3471851 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Arm/Group | Low Dose LY3471851 (Induction Treatment Period) | High Dose LY3471851 (Induction Treatment Period)
Number analyzed (Participants) | 26 | 26
microgram per milliliter (µg/mL) | 91.3 (49) | 139 (105)

ADVERSE EVENTS:
Time Frame: Baseline to Follow-up (Up To Week 58)
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | High Dose LY3471851 (Induction Treatment Period) | Low Dose LY3471851 (Induction Treatment Period) | Placebo (Induction Treatment Period) | High Dose LY3471851 (Maintenance Treatment Period) | Low Dose LY3471851 (Maintenance Treatment Period) | Placebo (Maintenance Treatment Period) | High Dose LY3471851 (Extension Treatment Period) | High Dose LY3471851 (Post-Treatment Follow-up Period) | Low Dose LY3471851 (Post-Treatment Follow-up Period) | Placebo (Post-Treatment Follow-up Period)
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/35 | 0/14 | 0/8 | 0/10 | 0/5 | 0/26 | 0/25 | 0/30 | 0/11
Serious Adverse Events (participants affected / at risk) | 2/32 | 0/35 | 0/14 | 0/8 | 1/10 | 0/5 | 0/26 | 0/25 | 1/30 | 0/11
Other Adverse Events (participants affected / at risk) | 20/32 | 15/35 | 5/14 | 4/8 | 6/10 | 1/5 | 5/26 | 0/25 | 1/30 | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose LY3471851 (Induction Treatment Period) (N=32) | Low Dose LY3471851 (Induction Treatment Period) (N=35) | Placebo (Induction Treatment Period) (N=14) | High Dose LY3471851 (Maintenance Treatment Period) (N=8) | Low Dose LY3471851 (Maintenance Treatment Period) (N=10) | Placebo (Maintenance Treatment Period) (N=5) | High Dose LY3471851 (Extension Treatment Period) (N=26) | High Dose LY3471851 (Post-Treatment Follow-up Period) (N=25) | Low Dose LY3471851 (Post-Treatment Follow-up Period) (N=30) | Placebo (Post-Treatment Follow-up Period) (N=11)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulval abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose LY3471851 (Induction Treatment Period) (N=32) | Low Dose LY3471851 (Induction Treatment Period) (N=35) | Placebo (Induction Treatment Period) (N=14) | High Dose LY3471851 (Maintenance Treatment Period) (N=8) | Low Dose LY3471851 (Maintenance Treatment Period) (N=10) | Placebo (Maintenance Treatment Period) (N=5) | High Dose LY3471851 (Extension Treatment Period) (N=26) | High Dose LY3471851 (Post-Treatment Follow-up Period) (N=25) | Low Dose LY3471851 (Post-Treatment Follow-up Period) (N=30) | Placebo (Post-Treatment Follow-up Period) (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site reaction (General disorders) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 8 (21) | 6 (20) | 0 (0) | 1 (12) | 0 (0) | 0 (0) | 2 (9) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 7 (9) | 2 (2) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (10) | 1 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 4 (11) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 3 (5) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT04677179/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/79/NCT04677179/SAP_001.pdf